CLINICAL TRIAL: NCT05797012
Title: The Association Among Headache Severity, Head Posture, Cervical Muscle Endurance, and Neck Disorders in Individuals With Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 83116987-711
Record Dates: First submitted 2023-03-16; First posted 2023-04-04 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Migraine Disorders
Keywords: Headache; Head posture; Neck disorders; Migraine; Cervical endurance
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals with migraine (Other): To assess headache severity, head posture, cervical muscle endurance and neck disorders.
  Interventions: Other: To assess headache severity, head posture, cervical muscle endurance and neck disorders.

INTERVENTIONS:
Other: To assess headache severity, head posture, cervical muscle endurance and neck disorders. — To assess headache severity, head posture, cervical muscle endurance and neck disorders.

SUMMARY:
To determine the relationship among headache severity, head posture, cervical muscle endurance and neck disorders in individuals with migraine.

DETAILED DESCRIPTION:
Headache is a general health problem that can be seen in different age groups, is common, depends on many factors, and has a lot of individual and socioeconomic effects. It is stated that the rate of individuals who experience a headache at least once in their lifetime is very high in the general population. Migraine is one of the most common types of primary headache. Neck pain and cervical dysfunctions in individuals with migraine have been the subject of many studies. It is seen that studies examining the relationship between cervical region musculoskeletal system disorders and headache in different types of headaches are increasing day by day. This study aims to determine the relationship among headache severity, head posture, cervical muscle endurance and neck disorders in individuals with migraine. In addition, the relationship between these parameters and quality of life will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with migraine at any time in his life and complaining of headache,
* Not having any diagnosed chronic disease,
* No past or present mental illness,
* Individuals who can speak, read and write Turkish.

Exclusion Criteria:

* Having any neurological, psychiatric or cognitive disorder,
* Individuals who cannot speak, read or write Turkish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Headache severity | 1 day
  Headache Impact Test-6 (HIT-6) will be used to question individuals' headache. This test, which consists of 6 items, evaluates the problems that arise due to headache in a wide framework. It provides information based on the patient's self-report. The HIT-6 score ranges from 36 to 78 points. A higher score indicates more influence. Turkish validity and reliability study of HIT-6 was conducted.
Head posture | 1 day
  Head posture will be recorded in degrees (°) by measuring the horizontal plane and the angle between the seventh cervical vertebra (C7) and the ear with an electrogoniometer (BASELINE® goniometer, Digital Absolute+Axis, Fabrication Enterprises (White Plains, New York)). None of the individuals will be informed about the head position to avoid bias in the study.
Cervical muscle endurance | 1 day
  The endurance of the cervical muscles will be evaluated with the deep cervical flexor endurance test and the cervical extensor endurance test.
Neck disorders | 1 day
  Neck disorders will be assessed by the Bournemouth Questionnaire (BQ) in 2002. BQ consists of 7 questions in total. Each question scores between 0 and 10. Although the highest score is 70, a high score indicates a high level of disability. The content of the questionnaire consists of variables that must be questioned for individuals with neck pain, such as pain severity, the effect of pain on activities of daily living and social life, anxiety-depression level, kinesiophobia, and coping with pain. The validity and reliability of the Turkish version of the BQ has been proven.
General quality of life | 1 day
  The Nottingham Health Profile (NHP) is a general quality of life questionnaire that measures a person's perceived health problems and the extent to which these problems affect normal daily activities. The questionnaire consists of 38 items. Questions are answered as 'yes' or 'no'. The questionnaire assesses six parameters related to health status. These parameters are; pain (8 items), physical activity (8 items), energy (3 items), sleep (5 items), social isolation (5 items), and emotional reactions (9 items). Each sub-parameter is scored between 0-100. 0 indicates best health, and 100 indicates worst health. The total NHP score is derived from the sum of the subscores.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Merkez, Tokat Province, Turkey (Türkiye)